CLINICAL TRIAL: NCT00593528
Title: Randomized Study With Medico-economic Evaluation Comparing the Use of PTFE Covered Stents vs Naked Stent in the TIPS (Transjugular Intra-hepatic Porto-systemic Shunt)
Brief Title: PTFE Covered Stents Versus Naked Stents in the TIPS (Transjugular Intra-hepatic Porto-systemic Shunt)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STIC07-JMP/TIPS-PTFE; 2007-A00857-46 (Other: EudraCT Number)
Record Dates: First submitted 2007-12-17; First posted 2008-01-15 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cirrhotic Portal Hypertension
Keywords: Cirrhosis, STIC TIPS, Portal Hypertension, Transjugular Intrahepatic Portosystemic Shunt , Stents, PTFE; cirrhotic HTP
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Naked Stents
  Interventions: Device: Naked Stents: Wallstent® (Boston Scientific), Luminexx® (Bard), Zilver® (Cook), Palmaz Genesis® and Smart Control® (Cordis); Procedure: Transjugular intrahepatic portosystemic shunt (TIPS)
- B (Experimental): PTFE Covered Stents
  Interventions: Device: PTFE Covered Stents: Fluency® (Bard), Advanta V12® (Atrium) and Viatorr® (Gore); Procedure: Transjugular intrahepatic portosystemic shunt (TIPS)

INTERVENTIONS:
Device: Naked Stents: Wallstent® (Boston Scientific), Luminexx® (Bard), Zilver® (Cook), Palmaz Genesis® and Smart Control® (Cordis) — Vascular Stents
  Arms: A
Device: PTFE Covered Stents: Fluency® (Bard), Advanta V12® (Atrium) and Viatorr® (Gore) — Vascular Stents
  Arms: B
Procedure: Transjugular intrahepatic portosystemic shunt (TIPS) — Transjugular intrahepatic portosystemic shunt (TIPS)

SUMMARY:
Transjugular intrahepatic portosystemic shunts (TIPS) have been increasingly used for the treatment of complications of portal hypertension in patients with cirrhosis.

The initial experiment of the TIPS was reported during the 1990s with stents of various brands, manufacture and sizes, but all "non covered", thus owing the pseudointimal hyperplasia growing inside the stent, which progressively decreases the diameter of the shunt and thus its efficacy. Since the beginning of the 2000s, appeared stents known as "covered" by polytetrafluoroethylene (PTFE) designed to reduce the obstruction rate and thus the frequency shunt revisions. However, these stents are, on average, 2.5 times more expensive than the non covered stents and the cost-effectiveness ratio of the TIPS according to the type of stents used has not been assessed.

The aim of this multicentric and randomized study is to assess the cost-effectiveness ratio of these 2 principles of TIPS, the one using stents covered by PTFE, relatively expensive but seldom becoming obstructed, and the other using non covered stents, less expensive than PTFE but requiring regular gestures of redilatation.

Population concerned: Patients with a cirrhotic portal hypertension responsible for:

* recurrent variceal bleeding
* refractory ascite (or hydrothorax)

ELIGIBILITY:
Inclusion Criteria:

* Presence of a cirrhosis as documented by previous liverbiopsy or typical clinical signs
* Indication validated of the TIPS (Bavéno IV), except not-controlled acute hemorrhagic :

  * Recurrent variceal bleeding after failure of the usual pharmacological and endoscopic methods
  * Refractory or recurrent ascites or difficult to treat
  * Refractory Hydrothorax

Exclusion Criteria:

* Non cirrhotic HTP
* CHILD C ≥12
* Complete portal vein thrombosis
* Usual contra-indication for TIPS :

  * Known or suspected Hepatocarcinoma by increase of the alpha-foetoprotein >100 UI/mL associated with the presence of at least one hepatic nodule
  * Cardiac insufficiency defined by a ventricular fraction of ejection < 40% with the echocardiography preliminary to the procedure
  * Pulmonary arterial hypertension (PAP > 40 mmHg)
  * Hepatic polycystosis
  * Intra-hepatic bile ducts dilatation,
  * Spontaneous clinical recurrent hepatic encephalopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-02-18 (Actual); Primary Completion 2011-07-11 (Actual); Study Completion 2011-07-11 (Actual)

PRIMARY OUTCOMES:
TIPS permeability rate | one year
Cost of the TIPS and patient care according to the type of stent used brought back to an indicator of effectiveness | one year

SECONDARY OUTCOMES:
Tolerance criteria : frequency of early complications like early thrombosis - probability of hepatic encephalopathy occurrence and gravity | one year
Quality of life | one year
Effectiveness criteria : survival rate - recurrence rate of the symptoms having justified the TIPS - various types of dysfunction | one year
Doppler : performance evaluation of Doppler for the diagnosis of dysfunction | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc PERARNAU, Doctor, Principal Investigator — CHRU TOURS
Locations (12):
- France (12):
  - Chru Bordeaux, Bordeaux
  - Chru Caen, Caen
  - Chru Clermont Ferrand, Clermont-Ferrand
  - Chru Dijon, Dijon
  - AP-HM / La Conception, Marseille
  - AP-HM / La Timone, Marseille
  - CHRU NANTES / Hôtel-Dieu, Nantes
  - CHRU NANTES / Hôpital Guillaume et René Laënnec, Nantes
  - Chru Nice, Nice
  - Chru Poitiers, Poitiers
  - CHRU de TOURS, Tours
  - Ap-Hp (Paul Brousse), Villejuif

REFERENCES:
- [Background] Perarnau JM, Noeldge G, Rossle M. [Intrahepatic portacaval anastomosis by the transjugular approach. Use of the Palmaz endoprosthesis]. Presse Med. 1991 Nov 9;20(36):1770-2. French. PMID 1836597
- [Background] Bureau C, Garcia-Pagan JC, Otal P, Pomier-Layrargues G, Chabbert V, Cortez C, Perreault P, Peron JM, Abraldes JG, Bouchard L, Bilbao JI, Bosch J, Rousseau H, Vinel JP. Improved clinical outcome using polytetrafluoroethylene-coated stents for TIPS: results of a randomized study. Gastroenterology. 2004 Feb;126(2):469-75. doi: 10.1053/j.gastro.2003.11.016. PMID 14762784
- [Background] Nishimine K, Saxon RR, Kichikawa K, Mendel-Hartvig J, Timmermans HA, Shim HJ, Uchida BT, Barton RE, Keller FS, Rosch J. Improved transjugular intrahepatic portosystemic shunt patency with PTFE-covered stent-grafts: experimental results in swine. Radiology. 1995 Aug;196(2):341-7. doi: 10.1148/radiology.196.2.7617843.
- [Background] Angermayr B, Cejna M, Koenig F, Karnel F, Hackl F, Gangl A, Peck-Radosavljevic M; Vienna TIPS Study Group. Survival in patients undergoing transjugular intrahepatic portosystemic shunt: ePTFE-covered stentgrafts versus bare stents. Hepatology. 2003 Oct;38(4):1043-50. doi: 10.1053/jhep.2003.50423. PMID 14512892
- [Background] Charon JP, Alaeddin FH, Pimpalwar SA, Fay DM, Olliff SP, Jackson RW, Edwards RD, Robertson IR, Rose JD, Moss JG. Results of a retrospective multicenter trial of the Viatorr expanded polytetrafluoroethylene-covered stent-graft for transjugular intrahepatic portosystemic shunt creation. J Vasc Interv Radiol. 2004 Nov;15(11):1219-30. doi: 10.1097/01.RVI.0000137434.19522.E5. PMID 15525740
- [Background] Barrio J, Ripoll C, Banares R, Echenagusia A, Catalina MV, Camunez F, Simo G, Santos L. Comparison of transjugular intrahepatic portosystemic shunt dysfunction in PTFE-covered stent-grafts versus bare stents. Eur J Radiol. 2005 Jul;55(1):120-4. doi: 10.1016/j.ejrad.2004.10.007. PMID 15950109
- [Background] Vignali C, Bargellini I, Grosso M, Passalacqua G, Maglione F, Pedrazzini F, Filauri P, Niola R, Cioni R, Petruzzi P. TIPS with expanded polytetrafluoroethylene-covered stent: results of an Italian multicenter study. AJR Am J Roentgenol. 2005 Aug;185(2):472-80. doi: 10.2214/ajr.185.2.01850472. PMID 16037523
- [Background] Rossle M, Siegerstetter V, Euringer W, Olschewski M, Kromeier J, Kurz K, Langer M. The use of a polytetrafluoroethylene-covered stent graft for transjugular intrahepatic portosystemic shunt (TIPS): Long-term follow-up of 100 patients. Acta Radiol. 2006 Sep;47(7):660-6. doi: 10.1080/02841850600806324. PMID 16950701
- [Background] Gandini R, Konda D, Simonetti G. Transjugular intrahepatic portosystemic shunt patency and clinical outcome in patients with Budd-Chiari syndrome: covered versus uncovered stents. Radiology. 2006 Oct;241(1):298-305. doi: 10.1148/radiol.2411050347. Epub 2006 Aug 14. PMID 16908675
- [Background] Tripathi D, Redhead D. Transjugular intrahepatic portosystemic stent-shunt: technical factors and new developments. Eur J Gastroenterol Hepatol. 2006 Nov;18(11):1127-33. doi: 10.1097/01.meg.0000236871.78280.a7. PMID 17033430
- [Background] Riggio O, Angeloni S, Nicolao F, Ridola L, Salvatori FM et al. Hepatic Encephalopathy is more frequent and severe after Transjugular intrahepatic portosystemeic Shunt (TIPS) with PTFE-coveted stent-grafts. Hepatology 2006;44, suppl 1, 232
- [Result] Perarnau JM, Le Gouge A, Nicolas C, d'Alteroche L, Borentain P, Saliba F, Minello A, Anty R, Chagneau-Derrode C, Bernard PH, Abergel A, Ollivier-Hourmand I, Gournay J, Ayoub J, Gaborit C, Rusch E, Giraudeau B; STIC-TIPS group. Covered vs. uncovered stents for transjugular intrahepatic portosystemic shunt: a randomized controlled trial. J Hepatol. 2014 May;60(5):962-8. doi: 10.1016/j.jhep.2014.01.015. Epub 2014 Jan 27. PMID 24480619